CLINICAL TRIAL: NCT02064985
Title: An Open Label, Single Centre, Randomised, Phase IV, Pharmacokinetic, Pharmacodynamic, and Safety Study to Evaluate Single and Multiple Doses of 45, 60, and 90 mg of Ticagrelor in Chinese Patients With Stable Coronary Heart Disease
Brief Title: Ticagrelor China Pharmacokinetic/Pharmacodynamic Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5130C00086
Record Dates: First submitted 2014-02-12; First posted 2014-02-17 (Estimated); Results first posted 2016-05-11 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-03

CONDITIONS: Stable Coronary Heart Disease (CHD)
MeSH Terms: interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ticagrelor 45mg (Experimental): A single dose of ticagrelor 45 mg on Day 1 followed by 45 mg twice daily (bid) on Days 3-6 and a 45mg single dose on Day 7.
  Interventions: Drug: Inhibition of Platelet Aggregation by "Brilinta"(Ticagrelor)
- Ticagrelor 60mg (Experimental): A single dose of ticagrelor 60 mg on Day 1 followed by 60 mg twice daily (bid) on Days 3-6 and a 60mg single dose on Day 7.
  Interventions: Drug: Inhibition of Platelet Aggregation by "Brilinta"(Ticagrelor)
- Ticagrelor 90mg (Experimental): A single dose of ticagrelor 90 mg on Day 1 followed by 90 mg twice daily (bid) on Days 3-6 and a 90mg single dose on Day 7.
  Interventions: Drug: Inhibition of Platelet Aggregation by "Brilinta"(Ticagrelor)

INTERVENTIONS:
Drug: Inhibition of Platelet Aggregation by "Brilinta"(Ticagrelor) — To determine the Inhibition of Platelet Aggregation (IPA) profiles of single and multiple doses of ticagrelor 45, 60, and 90 mg in Chinese patients with stable coronary heart disease (CHD) on chronic low dose ASA (75-100mg daily).
  Other Names: "Brilinta"(Ticagrelor)

SUMMARY:
open label, single centre, randomised, Phase IV, pharmacokinetic, pharmacodynamic, and safety study to evaluate single and multiple doses of 45, 60, and 90 mg of ticagrelor in Chinese patients with stable coronary heart disease

DETAILED DESCRIPTION:
Up to 36 patients will be randomized in order to ensure 10 patients per treatment are evaluable.Ticagrelor will be supplied as 45 mg, 60mg, and 90mg tablets. Following an 8 hour fast on single dose on Day 1 and Day 7; on multiple doses from Day 3 to Day 6. Prior to the first dose of study drug there will be a screening period of maximum of 19 days. Patients will report to the clinical pharmacology unit (CPU) on Day -2 and will remain confined there until completion of study procedures on Day 7, the patients will be discharged on Day 8. In addition, patients will return to the CPU for a follow up visit 2 to 5 days after the last dose. Each patients participation, including the screening period, will take approximately 33 days.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated written informed consent prior to any study specific procedures.
2. Female or male Chinese (as defined by Chinese Regulatory) patients aged 18 years or older with suitable veins for cannulations or repeated venipunctures.
3. Documented stable coronary heart disease (CHD) fulfilling all of the following, and taking 75-100 mg ASA daily treatment:

   Diagnosed stable angina pectoris per the guidance of Chinese Society of Cardiology published in 2007, patients with angina severity classified as I and II of Canadian Cardiovascular Society grading of angina pectoris.
4. Female patients without pregnant potential

Exclusion Criteria:

1. Any indication for oral anticoagulant or dual antiplatelet treatment and chronic ASA with doses greater than 100 mg/day.
2. Concomitant therapy with strong CYP3A inhibitors, CYP3A substrates with narrow therapeutic index, or strong CYP3A inducers within 14 days preceding the first dose of study medication and during study treatment.
3. Increased bleeding risk.
4. Contraindication or other reason that ASA or ticagrelor should not be administered
5. Patients that are scheduled for revascularization (eg, PCI, CABG) during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Li, PhD, Principal Investigator — The 3rd Hospital of Peking University
Locations (1):
- Research Site, Beijing, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was recruited on February 27th 2014 and the last patient's informed consent was obtained on Oct 24th 2014.
Pre-assignment Details: 22 participants did not meet includion/exclusion criteria. 2 participants withdrawed from study due to subject decision.1 participant withdrawed due to other reason. 36 participants were randomized and received study medication.
Period: Overall Study
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Started | 12 | 12 | 12
Completed | 12 | 12 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (9.8) | 61.3 (7.0) | 57.9 (12.6) | 59.5 (9.9)
Age, Customized [Number; unit: Participants]
  < 65 years | 9 | 8 | 8 | 25
  >=65 years | 3 | 4 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 8
  Male | 9 | 10 | 9 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 12 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 12 | 12 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: IPA on Day 1
Description: The Inhibition of Platelet Aggregation (IPA) profiles of single and multiple doses of ticagrelor 45, 60, and 90 mg in Chinese patients with stable coronary heart disease (CHD) on chronic low dose ASA (75-100mg daily).
  Primary variable: IPA (final extent) induced by 20µM ADP at each assessment point after single and multiple doses of ticagrelor measured by Light-Transmittance Aggregometry (LTA).
Time Frame: Baseline and at 0.5 hour, 1 hour, 2 hours, 3 hours, 6 hours, 12 hours, 24 hours, 36 hours,48 hours after dose intake on Day 1
Population: All randomly assigned patients who received at least 1 dose of ticagrelor with post-dose PD measurements available and no protocol deviation considered to significantly affect the integrity of PD results (eg, non-compliance with study drug).
Measure: Mean (Standard Deviation); unit: % IPA
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
% IPA
  0.5 hour after dose intake | 27.09 (25.956) | 25.87 (27.036) | 33.34 (31.238)
  1 hour after dose intake | 57.20 (26.563) | 50.97 (32.747) | 61.64 (31.244)
  2 hours after dose intake | 82.24 (21.160) | 84.10 (17.645) | 86.11 (22.213)
  3 hours after dose intake | 88.44 (11.786) | 90.18 (9.232) | 96.24 (6.396)
  6 hours after dose intake | 85.02 (8.965) | 94.32 (6.243) | 94.02 (6.190)
  12 hours after dose intake | 71.25 (16.518) | 85.70 (15.237) | 90.70 (8.117)
  24 hours after dose intake | 44.11 (34.165) | 49.38 (25.153) | 66.48 (21.200)
  36 hours after dose intake | 40.09 (28.211) | 46.23 (17.352) | 55.64 (29.446)
  48 hours after dose intake | 23.56 (22.956) | 27.25 (17.993) | 43.04 (25.178)

2. Secondary Outcome: Percent Change From Baseline in PRU on Day 1
Description: Percent Change from baseline in Platelet P2Y12 Reaction Units (PRU)(measured by VerifyNow) profiles of multiple doses of ticagrelor 45, 60, and 90 mg in Chinese patients with stable coronary heart disease on chronic low dose ASA.
Time Frame: as for outcome 1
Population: All randomized patients who received at least one dose of investigational product with post-dose PD measurements available and no protocol deviation considered to significantly affect the integrity of PD results (e.g., non-compliance with study drug) will be included in the PD analysis set.
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
% change from baseline
  0.5 hour after dose intake | -19.20 (13.712) | -13.76 (22.786) | -19.59 (23.880)
  1 hour after dose intake | -60.00 (27.295) | -35.25 (28.795) | -67.70 (30.613)
  2 hours after dose intake | -72.60 (16.492) | -61.23 (23.304) | -78.85 (18.775)
  3 hours after dose intake | -71.58 (22.220) | -75.42 (15.315) | -87.97 (11.134)
  6 hours after dose intake | -60.27 (25.208) | -67.98 (16.709) | -81.08 (11.024)
  12 hours after dose intake | -41.93 (23.584) | -47.15 (20.310) | -73.47 (13.705)
  24 hours after dose intake | -35.94 (20.706) | -28.34 (19.865) | -54.61 (19.553)
  36 hours after dose intake | -9.57 (17.655) | -1.91 (18.120) | -22.59 (24.694)
  48hours after dose intake | -15.19 (23.331) | -0.57 (13.070) | -16.38 (18.164)

3. Secondary Outcome: Pharmacokinetics Parameters of Ticagrelor on Day 7(1)
Description: Pharmacokinetics parameters of Ticagrelor on Day 7---Cmax
Time Frame: Plasma concentration was measured at Pre-dose, 0.5, 1, 2, 3, 6 and 12 hours post dose on Day 7
Population: All randomized patients who received at least one dose of investigational product with post-dose PK measurements available and no protocol deviation considered to significantly affect PK of ticagrelor and its metabolite, AR C124910XX, will be included in the PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
ng/mL | 616.0 (37.09) | 689.4 (33.64) | 1273 (43.00)

4. Secondary Outcome: Safety---Vital Signs Over Time---Blood Pressure
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Vital signs (seated blood pressure [BP])
Time Frame: Baseline, Day 1 to Day 7 and 2 to 5 days after last dose
Population: All patients who receive at least one administration of the investigational product and for whom any post-dose data are available will be included in the safety analysis set.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
mmHg
  Diastolic Blood Pressure- Baseline | 84.6 (7.6) | 77.1 (9.7) | 74.8 (15.5)
  Diastolic Blood Pressure- Day 1 | 85.3 (9.0) | 78.2 (9.6) | 74.6 (11.3)
  Diastolic Blood Pressure-Day 2 | 82.3 (9.3) | 74.8 (7.5) | 74.2 (11.3)
  Diastolic Blood Pressure-Day 3 | 79.2 (11.0) | 75.2 (7.5) | 74.3 (11.5)
  Diastolic Blood Pressure-Day 4 | 80.7 (11.4) | 78.2 (8.7) | 73.3 (11.2)
  Diastolic Blood Pressure-Day 5 | 80.8 (10.3) | 75.2 (5.6) | 74.7 (9.5)
  Diastolic Blood Pressure-Day 6 | 79.8 (8.7) | 77.4 (4.8) | 73.9 (11.5)
  Diastolic Blood Pressure-Day 7 | 80.8 (7.7) | 75.6 (6.7) | 74.0 (11.5)
  Diastolic Blood Pressure-2-5 days after last Dose | 80.3 (6.8) | 74.7 (6.7) | 71.3 (9.2)
  Systolic Blood Pressure (mmHg)-Baseline | 134.6 (14.6) | 129.2 (11.6) | 132.1 (14.5)
  Systolic Blood Pressure-Day 1 | 132.2 (12.0) | 135.7 (19.2) | 127.4 (11.9)
  Systolic Blood Pressure-Day 2 | 130.3 (15.0) | 131.4 (20.0) | 123.1 (14.2)
  Systolic Blood Pressure-Day 3 | 128.3 (11.0) | 130.1 (18.8) | 123.8 (9.5)
  Systolic Blood Pressure-Day 4 | 131.3 (12.8) | 132.8 (15.3) | 126.1 (12.0)
  Systolic Blood Pressure-Day 5 | 129.4 (11.0) | 131.3 (18.6) | 125.1 (11.0)
  Systolic Blood Pressure-Day 6 | 126.8 (14.0) | 133.5 (19.5) | 119.1 (9.2)
  Systolic Blood Pressure-Day 7 | 128.9 (11.8) | 129.4 (22.7) | 122.1 (11.3)
  Systolic Blood Pressure-2-5 days after last Dose | 126.0 (16.0) | 132.3 (17.3) | 124.7 (13.9)

5. Primary Outcome: IPA on Day 7
Description: as for outcome 1
Time Frame: Baseline and at 0 hour, 0.5 hour, 1 hour, 2 hours, 3 hours, 6 hours, 12 hours after dose intake on Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % IPA
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
% IPA
  0 hour after dose intake | 79.69 (20.547) | 89.26 (7.857) | 95.10 (6.910)
  0.5 hour after dose intake | 84.70 (15.998) | 89.96 (7.985) | 96.90 (3.602)
  1 hour after dose intake | 88.82 (15.639) | 93.28 (7.589) | 96.47 (4.184)
  2 hours after dose intake | 88.30 (17.325) | 94.62 (3.787) | 98.29 (3.526)
  3 hours after dose intake | 91.00 (13.212) | 97.01 (2.258) | 98.86 (2.664)
  6 hours after dose intake | 91.13 (14.344) | 92.94 (17.847) | 98.87 (2.598)
  12 hours after dose intake | 86.55 (16.918) | 92.01 (7.316) | 96.81 (4.219)

6. Secondary Outcome: Percent Change From Baseline in PRU on Day 7
Description: as for outcome 2
Time Frame: Baseline and at 0 hour, 0.5 hour, 1 hour, 2 hours, 3 hours, 6 hours, 12 hours after dose intake on Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % change from baseline
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
% change from baseline
  0.5 hour after dose intake | -77.90 (17.632) | -80.07 (14.691) | -89.33 (8.923)
  1 hour after dose intake | -79.70 (17.742) | -78.40 (18.103) | -94.10 (6.746)
  2 hours after dose intake | -82.23 (17.304) | -85.00 (12.020) | -88.81 (13.595)
  3 hours after dose intake | -79.98 (18.434) | -86.96 (12.868) | -92.13 (9.288)
  6 hours after dose intake | -76.71 (20.067) | -75.07 (14.806) | -91.48 (7.928)
  12 hours after dose intake | -63.63 (23.767) | -69.03 (19.867) | -88.60 (8.816)

7. Secondary Outcome: TIPA(Max)---Day 1
Description: The time to peak IPA (TIPAmax) was estimated for ADP-induced final extent IPA.
Time Frame: Day 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
hour | 3.0 (17.632) [2.5 to 6.0] | 4.5 (14.691) [3.0 to 6.0] | 2.5 (8.923) [2.0 to 3.0]

8. Secondary Outcome: TIPA(Max)---Day 7
Description: The time to peak IPA (TIPAmax) was estimated for ADP-induced final extent IPA.
Time Frame: Day 7
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
hour | 1.5 (17.632) [1.0 to 4.5] | 6.0 (14.691) [1.8 to 6.0] | 1.3 (8.923) [0.0 to 2.5]

9. Secondary Outcome: AUEC(Final Extent) on Day 1
Description: The area-under-the-effect curve (AUEC) was estimated for ADP-induced final extent IPA.
Time Frame: IPA was measured at Pre-dose, 0.5, 1, 2, 3, 6, 12, 24, 36, and 48 hours post dose on Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: %*h
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
%*h | 2474.4 (949.3) [1.0 to 4.5] | 2819.4 (707.17) [1.8 to 6.0] | 3301.0 (788.72) [0.0 to 2.5]

10. Secondary Outcome: AUEC(Final Extent) on Day 7
Description: The area-under-the-effect curve (AUEC) was estimated for ADP-induced final extent IPA.
Time Frame: IPA was measured at Pre-dose, 0.5, 1, 2, 3, 6 and 12 hours post dose on Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: %*h
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
%*h | 1069.9 (176.89) [1.0 to 4.5] | 1120.1 (108.44) [1.8 to 6.0] | 1176.9 (33.03) [0.0 to 2.5]

11. Secondary Outcome: Pharmacokinetics Parameters of Ticagrelor on Day 1(3)
Description: The pharmacokinetics parameter of ticagrelor on Day 1---tmax and t1/2
Time Frame: Plasma concentration was measured at Pre-dose, 0.5, 1, 2, 3, 6, 12, 24, 36, and 48 hours post dose on Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
hour
  tmax | 2.00 (38.02) [1.00 to 2.00] | 3.00 (34.14) [1.00 to 6.00] | 2.00 (37.39) [1.00 to 3.03]
  t½ | 10.07 (51.42) [9.21 to 15.9] | 9.008 (32.46) [7.94 to 12.5] | 9.802 (53.84) [7.81 to 13.7]

12. Secondary Outcome: Pharmacokinetics Parameters of Ticagrelor on Day 1(2)
Description: The pharmacokinetics parameters of Ticagrelor on Day 1---AUC(0-inf), AUC(0-12h) and AUC(0-t).
Time Frame: Plasma concentration was measured at Pre-dose, 0.5, 1, 2, 3, 6, 12, 24, 36, and 48 hours post dose on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
h*ng/mL
  AUC(0-inf) | 3220 (51.42) | 3633 (32.46) | 6234 (53.84)
  AUC(0-t) | 3102 (49.79) | 3533 (31.68) | 6017 (51.71)
  AUC(0-12h) | 2114 (41.97) | 2313 (30.10) | 3983 (41.93)

13. Secondary Outcome: Pharmacokinetics Parameters of Ticagrelor on Day 7(2)
Description: The pharmacokinetics parameters of ticagrelor on Day 7---tmax
Time Frame: Plasma concentration was measured at Pre-dose, 0.5, 1, 2, 3, 6 and 12 hours post dose on Day 7
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
hour | 2.00 (37.09) [1.00 to 3.03] | 2.00 (33.64) [1.00 to 3.00] | 2.00 (43.00) [1.00 to 3.00]

14. Secondary Outcome: Pharmacokinetics Parameters of Metabolite (AR-C124910XX) on Day 1(1)
Description: Pharmacokinetics parameters of AR-C124910XX (active metabolite) on Day 1---Cmax
Time Frame: Plasma concentration was measured at Pre-dose, 0.5, 1, 2, 3, 6, 12, 24, 36, and 48 hours post dose on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
ng/mL | 88.28 (24.58) | 77.11 (53.92) | 138.6 (38.37)

15. Secondary Outcome: Pharmacokinetics Parameters of Metabolite (AR-C124910XX) on Day 1(3)
Description: Pharmacokinetics parameters of AR-C124910XX (active metabolite) on Day 1: tmax and t1/2
Time Frame: Plasma concentration was measured at Pre-dose, 0.5, 1, 2, 3, 6, 12, 24, 36, and 48 hours post dose on Day 1
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
hour
  tmax | 2.00 (38.02) [2.00 to 3.00] | 3.00 (34.14) [2.00 to 6.00] | 3.00 (37.39) [2.00 to 3.03]
  t½ | 13.16 (51.42) [8.22 to 17.1] | 11.64 (32.46) [8.00 to 20.0] | 11.29 (53.84) [8.74 to 21.5]

16. Secondary Outcome: Pharmacokinetics Parameters of Metabolite (AR-C124910XX) on Day 7(1)
Description: Pharmacokinetics parameters of Metabolite (AR-C124910XX) on Day 7---Cmax
Time Frame: Plasma concentration was measured at Pre-dose, 0.5, 1, 2, 3, 6 and 12 hours post dose on Day 7
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
ng/mL | 143.7 (26.32) | 180.1 (49.83) | 300.6 (31.74)

17. Secondary Outcome: Pharmacokinetics Parameters of Metabolite (AR-C124910XX) on Day 7(4)
Description: Pharmacokinetics parameters of AR-C124910XX (active metabolite) on Day 7---tmax
Time Frame: Plasma concentration was measured at Pre-dose, 0.5, 1, 2, 3, 6 and 12 hours post dose on Day 7
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
hour | 2.00 (38.02) [2.00 to 6.00] | 2.00 (34.14) [2.00 to 3.00] | 2.54 (37.39) [2.00 to 3.10]

18. Secondary Outcome: Pharmacokinetics Parameters of Metabolite : Parent on Day 1--Cmax
Description: To determine Cmax ratio for the metabolite to that of the parent compound on Day 1
Time Frame: Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
ratio | 0.2277 (0.08984) [2.00 to 6.00] | 0.2146 (0.06333) [2.00 to 3.00] | 0.2005 (0.08334) [2.00 to 3.10]

19. Secondary Outcome: Pharmacokinetics Parameters of Metabolite : Parent on Day 7---Cmax
Description: To determine Cmax ratio of metabolite to that of the parent compound on Day 7
Time Frame: Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
ratio | 0.2657 (0.07820) [2.00 to 6.00] | 0.3082 (0.1223) [2.00 to 3.00] | 0.2646 (0.06758) [2.00 to 3.10]

20. Secondary Outcome: Safety---Physical Examination, Summary of Abnormalities
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Physical examination
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
Participants
  Number of patients with abnormality | 5 (7.6) | 3 (9.7) | 2 (15.6)
  Abdomen | 1 (9.0) | 0 (9.6) | 0 (11.3)
  Cardiovascular | 0 (16.0) | 0 (17.3) | 0 (13.9)
  General appearance | 0 | 0 | 0
  Head and neck | 0 | 0 | 0
  Lymph nodes | 0 | 0 | 0
  Musculoskeletal / Extremities | 0 | 0 | 0
  Neurological | 0 | 0 | 0
  Respiratory | 0 | 0 | 0
  Skin | 4 | 3 | 2
  Thyroid | 0 | 0 | 0

21. Secondary Outcome: Safety---Hematology Laboratory Variables Over Time---hematocrit
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Haematology---hematocrit
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
ratio | 0.4083 (0.0365) | 0.4020 (0.0465) | 0.4153 (0.0369)

22. Secondary Outcome: Safety---All Allowed Concomitant Medications During Study Treatment
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Concomitant medications
Time Frame: All allowed concomitant medications during study treatment(up to 2-5 days after last dose), includes medications that began prior to randomization but were ongoing after randomization.
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
Participants
  Number of patients with allowed concomitant med | 12 (3.65) | 12 (1.86) | 12 (1.19)
  HMG CoA reductase inhibitors | 11 (0.297) | 12 (0.186) | 12 (0.216)
  ATORVASTATIN | 5 (0.200) | 8 (0.134) | 5 (0.109)
  SIMVASTATIN | 3 (0.301) | 4 (0.111) | 3 (0.179)
  ROSUVASTATIN | 3 (12.25) | 0 (17.89) | 4 (13.48)
  Beta blocking agents, selective | 9 (4.36) | 10 (5.91) | 6 (9.67)
  METOPROLOL | 6 (1.5) | 6 (1.4) | 5 (2.6)
  BISOPROLOL | 3 (0.36) | 5 (0.33) | 1 (0.25)
  ACE inhibitors, plain | 5 (1.6) | 2 (2.0) | 6 (2.5)
  PERINDOPRIL | 2 | 0 | 3
  FOSINOPRIL | 1 | 1 | 2
  ENALAPRIL | 0 | 1 | 1
  BENAZEPRIL | 1 | 0 | 0
  IMIDAPRIL | 1 | 0 | 0
  Dihydropyridine derivatives | 4 | 3 | 2
  AMLODIPINE | 3 | 3 | 2
  NIFEDIPINE | 1 | 0 | 0
  Other cardiac preparations | 4 | 2 | 2
  TRIMETAZIDINE | 4 | 2 | 1
  TRIMETAZIDINE HYDROCHLORIDE | 0 | 0 | 1
  Biguanides | 3 | 2 | 2
  METFORMIN | 2 | 2 | 2
  METFORMIN HYDROCHLORIDE | 1 | 0 | 0
  Organic nitrates | 1 | 2 | 3
  ISOSORBIDE MONONITRATE | 1 | 2 | 3
  Angiotensin II antagonists, plain | 3 | 1 | 1
  IRBESARTAN | 2 | 1 | 0
  LOSARTAN | 1 | 0 | 0
  TELMISARTAN | 0 | 0 | 1
  Alpha glucosidase inhibitors | 3 | 1 | 0
  ACARBOSE | 3 | 1 | 0
  Insulins and analogues for injection, fast-acting | 1 | 3 | 0
  INSULIN | 1 | 2 | 0
  INSULIN HUMAN | 0 | 1 | 0
  Enzymes | 0 | 1 | 2
  KALLIDINOGENASE | 0 | 1 | 2
  Folic acid and derivatives | 2 | 1 | 0
  FOLIC ACID | 2 | 1 | 0
  Alpha and beta blocking agents | 1 | 0 | 1
  CARVEDILOL | 1 | 0 | 1
  Other therapeutic products | 0 | 2 | 0
  CHINESE TRADITIONAL MEDICINE NOS | 0 | 1 | 0
  HERBAL NOS | 0 | 1 | 0
  Preparations inhibiting uric acid production | 2 | 0 | 0
  ALLOPURINOL | 2 | 0 | 0
  Sulfonamides, urea derivatives | 1 | 0 | 1
  GLIMEPIRIDE | 0 | 0 | 1
  GLIQUIDONE | 1 | 0 | 0
  ANTIHYPERTENSIVES | 0 | 0 | 1
  ANTIHYPERTENSIVES | 0 | 0 | 1
  Aldose reductase inhibitors | 0 | 1 | 0
  EPALRESTAT | 0 | 1 | 0
  Angiotensin II antagonists and diuretics | 0 | 0 | 1
  HYDROCHLOROTHIAZIDE+ LOSARTAN | 0 | 0 | 1
  Antidepressants in combination with psycholeptics | 0 | 1 | 0
  FLUPENTIXOL+MELITRACEN | 0 | 1 | 0
  Benzodiazepine derivatives | 0 | 1 | 0
  ESTAZOLAM | 0 | 1 | 0
  Benzothiazepine derivatives | 1 | 0 | 0
  DILTIAZEM | 1 | 0 | 0
  Comb/complexes aluminium, calcium, magnesium comps | 1 | 0 | 0
  HYDROTALCITE | 1 | 0 | 0
  Fibrates | 0 | 0 | 1
  FENOFIBRATE | 0 | 0 | 1
  Insulins and analogues for inj,intermediate-acting | 1 | 0 | 0
  HUMULIN 70/30 | 1 | 0 | 0
  Insulins/analogues for inj,int/long-act+fast-actin | 1 | 0 | 0
  INSULIN ASPART | 1 | 0 | 0
  Nicotinic acid and derivatives | 0 | 1 | 0
  ACIPIMOX | 0 | 1 | 0
  Other antifungals for topical use | 1 | 0 | 0
  TERBINAFINE HYDROCHLORIDE | 1 | 0 | 0
  Other drugs for peptic ulcer and GORD | 0 | 0 | 1
  GEFARNATE | 0 | 0 | 1
  Other vasodilators used in cardiac diseases | 0 | 1 | 0
  NICORANDIL | 0 | 1 | 0
  Thiazolidinediones | 0 | 1 | 0
  ROSIGLITAZONE | 0 | 1 | 0

23. Secondary Outcome: Safety---Causally Related Adverse Events by System Organ Class and Preferred Term
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Assessment of adverse events
Time Frame: Includes adverse events with an onset date on or after the date of first dose and up to and including the last study visit (up to 2-5 days after last dose).
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
Participants
  Patients with any causally related AE | 1 (3.65) | 2 (1.86) | 2 (1.19)
  Respiratory, thoracic and mediastinal disorders | 0 (0.297) | 2 (0.186) | 2 (0.216)
  Dyspnoea | 0 (0.200) | 2 (0.134) | 1 (0.109)
  Haemoptysis | 0 (0.301) | 0 (0.111) | 1 (0.179)
  Gastrointestinal disorders | 1 (12.25) | 0 (17.89) | 0 (13.48)
  Diarrhoea | 1 (4.36) | 0 (5.91) | 0 (9.67)
  Investigations | 1 (1.5) | 0 (1.4) | 0 (2.6)
  Occult blood positive | 1 (0.36) | 0 (0.33) | 0 (0.25)

24. Secondary Outcome: Pharmacokinetics Parameters of Ticagrelor on Day 1(1)
Description: The pharmacokinetics parameters of Ticagrelor on Day 1---Cmax
Time Frame: Plasma concentration was measured at Pre-dose, 0.5, 1, 2, 3, 6, 12, 24, 36, and 48 hours post dose on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
ng/mL | 464.0 (38.02) | 413.9 (34.14) | 822.1 (37.39)

25. Secondary Outcome: Pharmacokinetics Parameters of Ticagrelor on Day 7(3)
Description: Pharmacokinetics parameters of Ticagrelor on Day 7---AUC(0-12h)
Time Frame: Plasma concentration was measured at Pre-dose, 0.5, 1, 2, 3, 6 and 12 hours post dose on Day 7
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
h*ng/mL | 3882 (41.67) | 4351 (36.74) | 8206 (50.92)

26. Secondary Outcome: Pharmacokinetics Parameters of Ticagrelor on Day 7(4)
Description: Pharmacokinetics parameters of Ticagrelor on Day 7---Accumulation ratio(ratio of Day 7 AUC(0-12h) to Day 1 AUC(0-12h))
Time Frame: Plasma concentration was measured at Pre-dose, 0.5, 1, 2, 3, 6 and 12 hours post dose on Day 7
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
ratio | 1.837 (23.57) | 1.882 (20.72) | 2.060 (22.84)

27. Secondary Outcome: Safety---Vital Signs Over Time---Height
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Vital signs (Height)
Time Frame: Baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
cm | 166.9 (7.6) | 168.8 (8.0) | 166.5 (7.7)

28. Secondary Outcome: Safety---Vital Signs Over Time---Weight
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Vital signs (Weight)
Time Frame: Baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
kg | 78.7 (10.2) | 73.8 (8.5) | 73.4 (9.8)

29. Secondary Outcome: Safety---Vital Signs Over Time---Pulse Rate
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Vital signs (Pulse Rate)
Time Frame: Baseline, Day 1 to Day 7 and 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: BEATS/MIN
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
BEATS/MIN
  Pulse Rate (BEATS/MIN)- Baseline | 63.3 (8.6) | 60.5 (6.8) | 59.1 (5.5)
  Pulse Rate (BEATS/MIN)- Day 1 | 64.2 (8.4) | 60.6 (6.5) | 61.3 (5.2)
  Pulse Rate (BEATS/MIN)- Day 2 | 64.6 (10.6) | 59.8 (7.3) | 63.3 (7.2)
  Pulse Rate (BEATS/MIN)- Day 3 | 67.3 (9.8) | 60.4 (7.1) | 61.3 (4.4)
  Pulse Rate (BEATS/MIN)- Day 4 | 65.3 (9.2) | 61.7 (5.5) | 63.7 (6.5)
  Pulse Rate (BEATS/MIN)- Day 5 | 66.7 (8.5) | 62.7 (7.1) | 64.2 (5.9)
  Pulse Rate (BEATS/MIN)- Day 6 | 66.8 (8.5) | 59.9 (7.2) | 64.1 (4.4)
  Pulse Rate (BEATS/MIN)- Day 7 | 65.4 (6.2) | 62.7 (7.8) | 62.9 (5.7)
  Pulse Rate(BEATS/MIN)- 2 to 5 days after last dose | 64.6 (10.9) | 61.8 (5.5) | 63.0 (6.8)

30. Secondary Outcome: Pharmacokinetics Parameters of Metabolite (AR-C124910XX) on Day 1(2)
Description: Pharmacokinetics parameters of AR-C124910XX (active metabolite) on Day 1---AUC(0-12h), AUC(0-t) and AUC(0-inf)
Time Frame: Plasma concentration was measured at Pre-dose, 0.5, 1, 2, 3, 6, 12, 24, 36, and 48 hours post dose on Day 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
h*ng/mL
  AUC(0-inf) | 921.5 (28.66) | 1108 (34.83) | 1644 (30.83)
  AUC(0-t) | 839.6 (25.23) | 906.0 (56.84) | 1534 (28.88)
  AUC(0-12h) | 464.0 (19.11) | 504.1 (55.41) | 835.9 (29.59)

31. Secondary Outcome: Pharmacokinetics Parameters of Metabolite (AR-C124910XX) on Day 7(2)
Description: Pharmacokinetics parameters of Metabolite (AR-C124910XX) on Day 7---AUC(0-12h)
Time Frame: Plasma concentration was measured at Pre-dose, 0.5, 1, 2, 3, 6 and 12 hours post dose on Day 7
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
h*ng/mL | 1069 (24.89) | 1314 (41.02) | 2254 (37.02)

32. Secondary Outcome: Pharmacokinetics Parameters of Metabolite (AR-C124910XX) on Day 7(3)
Description: Pharmacokinetics parameters of Metabolite (AR-C124910XX) on Day 7---Accumulation ratio(ratio of Day 7 AUC(0-12h) to Day 1 AUC(0-12h))
Time Frame: Plasma concentration was measured at Pre-dose, 0.5, 1, 2, 3, 6 and 12 hours post dose on Day 7
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
ratio | 2.304 (24.70) | 2.606 (28.34) | 2.697 (27.42)

33. Secondary Outcome: Safety---Hematology Laboratory Variables Over Time---Erythrocytes
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Haematology---Erythrocytes
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 10^12/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
10^12/L | 4.417 (0.319) | 4.409 (0.400) | 4.487 (0.427)

34. Secondary Outcome: Safety---Hematology Laboratory Variables Over Time---Hemoglobin
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Haematology---Hemoglobin
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
g/L | 137.3 (11.6) | 135.4 (15.2) | 138.6 (12.9)

35. Secondary Outcome: Safety---Hematology Laboratory Variables Over Time---Leukocytes
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Haematology---Leukocytes
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
10^9/L | 6.64 (1.23) | 6.30 (1.12) | 6.74 (1.29)

36. Secondary Outcome: Safety---Hematology Laboratory Variables Over Time---Platelets
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Haematology---Platelets
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
10^9/L | 205.3 (34.5) | 186.7 (38.5) | 227.3 (42.4)

37. Secondary Outcome: Safety---Clinical Chemistry Variables Over Time---Glucose
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Clinical Chemistry---Glucose
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
mmol/L | 7.48 (3.65) | 7.26 (1.86) | 5.78 (1.19)

38. Secondary Outcome: Safety---Clinical Chemistry Variables Over Time---Alanine Aminotransferase
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Clinical Chemistry---Alanine Aminotransferase
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ukat/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
ukat/L | 0.524 (0.297) | 0.429 (0.186) | 0.465 (0.216)

39. Secondary Outcome: Safety---Clinical Chemistry Variables Over Time---Aspartate Aminotransferase
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Clinical Chemistry---Aspartate Aminotransferase
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ukat/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
ukat/L | 0.497 (0.200) | 0.410 (0.134) | 0.433 (0.109)

40. Secondary Outcome: Safety---Clinical Chemistry Variables Over Time---Alkaline Phosphatase
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Clinical Chemistry---Alkaline Phosphatase
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ukat/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
ukat/L | 1.172 (0.301) | 1.027 (0.111) | 1.028 (0.179)

41. Secondary Outcome: Safety---Clinical Chemistry Variables Over Time---Creatinine
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Clinical Chemistry---Creatinine
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
umol/L | 81.92 (12.25) | 87.50 (17.89) | 83.50 (13.48)

42. Secondary Outcome: Safety---Clinical Chemistry Variables Over Time---Total Bilirubin
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Clinical Chemistry---Total Bilirubin
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
umol/L | 13.98 (4.36) | 14.58 (5.91) | 14.81 (9.67)

43. Secondary Outcome: Safety---Clinical Chemistry Variables Over Time---Sodium
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Clinical Chemistry---Sodium
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
mmol/L | 140.7 (1.5) | 140.8 (1.4) | 141.3 (2.6)

44. Secondary Outcome: Safety---Clinical Chemistry Variables Over Time---Potassium
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Clinical Chemistry---Potassium
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
mmol/L | 4.41 (0.36) | 4.47 (0.33) | 4.26 (0.25)

45. Secondary Outcome: Safety---Clinical Chemistry Variables Over Time---Chloride
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Clinical Chemistry---Chloride
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
mmol/L | 103.2 (1.6) | 103.9 (2.0) | 104.4 (2.5)

46. Secondary Outcome: Safety---Clinical Chemistry Variables Over Time---Phosphate
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Clinical Chemistry---Phosphate
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
mmol/L | 1.188 (0.183) | 1.154 (0.158) | 1.145 (0.101)

47. Secondary Outcome: Safety---Clinical Chemistry Variables Over Time---Albumin
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Clinical Chemistry---Albumin
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
g/L | 44.77 (1.51) | 44.68 (2.54) | 46.07 (2.25)

48. Secondary Outcome: Safety---Clinical Chemistry Variables Over Time---Protein
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Clinical Chemistry---Protein
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
g/L | 70.2 (3.6) | 69.8 (3.0) | 70.2 (4.5)

49. Secondary Outcome: Safety---Clinical Chemistry Variables Over Time---Blood Urea Nitrogen
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Clinical Chemistry---Blood Urea Nitrogen
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
mmol/L | 5.875 (1.500) | 6.392 (1.648) | 6.108 (1.366)

50. Secondary Outcome: Safety---Clinical Chemistry Variables Over Time---Bicarbonate
Description: The safety of ticagrelor in Chinese patients with stable coronary heart disease on chronic low dose ASA.
  Safety will be assessed by:
  • Clinical Chemistry---Bicarbonate
Time Frame: 2 to 5 days after last dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
mmol/L | 28.92 (2.77) | 28.55 (1.95) | 28.15 (3.20)

51. Secondary Outcome: Pharmacokinetics Parameters of Metabolite : Parent on Day 1--AUC(0-inf)
Description: To determine AUC(0-inf) ratio for the metabolite to that of the parent compound on Day 1
Time Frame: Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
ratio | 0.3310 (0.09838) | 0.3403 (0.07381) | 0.3106 (0.1283)

52. Secondary Outcome: Pharmacokinetics Parameters of Metabolite : Parent on Day 7---AUC(0-12h)
Description: To determine AUC(0-12h) ratio of metabolite to that of the parent compound on Day 7.
Time Frame: Day 7
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Number analyzed (Participants) | 12 | 12 | 12
ratio | 0.3132 (0.08899) | 0.3549 (0.1351) | 0.3153 (0.1120)

ADVERSE EVENTS:
Arm/Group | Ticagrelor 45mg | Ticagrelor 60mg | Ticagrelor 90mg
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 4/12 | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ticagrelor 45mg (N=12) | Ticagrelor 60mg (N=12) | Ticagrelor 90mg (N=12)
Tinea pedis (Infections and infestations) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Cardiac discomfort (Cardiac disorders) | 0 | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Occult blood positive (Investigations) | 1 | 0 | 0
Electrocardiogram ST-T change (Investigations) | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Principal Investigator may use the Study results (data generated at the site) and shall not publish or present any such results until the earlier of (i) the date of the first Study results publication and (ii) the end of the eighteen (18) month period following the completion, or early termination, of the Study at all participating sites.